CLINICAL TRIAL: NCT00186992
Title: Image Guided Radiotherapy for the Treatment of Musculoskeletal Tumors: A Phase II Prospective Evaluation of Radiation-related Treatment Effects
Brief Title: Radiation Therapy to Treat Musculoskeletal Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Lance Armstrong Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTSARC; NCI-2011-01222 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma, Ewing's; Rhabdomyosarcoma; Soft Tissue Sarcoma; Musculoskeletal Tumors
Keywords: Sarcoma; radiation therapy; Other musculoskeletal tumors
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Other): Eligible patients will be accessioned at the time of irradiation and undergo a pre-radiotherapy evaluation, treatment planning, image-guided radiotherapy delivery and intra-and post-irradiation evaluations.
  Interventions: Radiation: image-guided radiotherapy

INTERVENTIONS:
Radiation: image-guided radiotherapy — Conformal limited image radiotherapy is radiation therapy that targets tumors with a prescribed dose of radiation which allows the surrounding normal tissues to remain basically untreated.

SUMMARY:
Researchers at St. Jude Children's Research Hospital are looking for more effective ways to deliver radiation therapy to pediatric tumors of the bone and soft tissues. The goal of the study is to improve local control of musculoskeletal tumors with image-guided radiation therapy (IGRT) while minimizing radiation related side effects. IGRT uses computed tomography (CT), magnetic resonance imaging (MRI) and positron emission tomography (PET) images to precisely define tumor location and to carefully plan radiation treatment. This approach allows doctors to deliver highly conformal radiation therapy to the tumor while protecting nearby healthy normal tissues.

DETAILED DESCRIPTION:
The study focuses on the following primary Objectives:

* To estimate local control rates with image guided radiation therapy as defined in this study for patients with primary musculoskeletal tumors (MST).

  * Prospectively establish a baseline estimate of local control for patients with MST (Ewing's sarcoma family of tumors (ESFT), rhabdomyosarcoma (RMS) and non-rhabdomyosarcoma soft tissue sarcoma (STS)) treated with image guided radiation therapy.
  * Demonstrate that the increased level of conformality afforded by image guided radiation therapy does not reduce its efficacy relative to previously utilized non-image guided radiation therapy techniques in patients with Ewing's sarcoma family of tumors, resected soft tissue sarcomas, and group III rhabdomyosarcomas.
  * Assess local and regional patterns of failure for patients with MST treated with image guided radiation therapy relative to their targeted volumes.
  * Provide a long term (>5 year) estimate of local disease control for patients with MST (Ewing's sarcoma family of tumors (ESFT)), rhabdomyosarcoma (RMS), and non-rhabdomyosarcoma soft tissue sarcoma (STS) treated with image guided radiation therapy.

The study focuses on the following secondary objectives:

* Establish a quantitative baseline estimate of radiation dose-related changes in normal tissues using novel objective measures of somatic change, musculoskeletal function, tissue biochemistry and physiology.

  o Investigate the dose and volume relationship for the developing physis and cortical bone using physical measures and imaging evaluations including:
  * Prospectively investigate whether an age based radiotherapeutic threshold of dose and volume that will induce premature physis closure and alter long bone length can be quantitatively identified.
  * Quantitatively explore the impact of radiation on cortical bone thinning and long bone curvature.
  * Relate radiation dose and volume to late (10+ year) alterations in bone integrity.
* Describe the severity and time course of radiation-induced changes in the soft tissues including muscle.

  * Delineate sequential changes in muscular volume, muscle function and organ function (delineated by imaging and measures of physical function) following image guided radiation for specific muscular groups.
  * Correlate the temporal changes in muscular volume and function with changes in vascularity and metabolism defined by imaging studies.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 25 years (new enrollments only). No age limit on participants who reconsent or reenroll.
* Musculoskeletal tumor involving the primary site of origin requiring definitive, pre-operative or post-operative irradiation to that primary site.
* No prior therapeutic irradiation at the primary site except for emergent radiation to the primary site lasting 1 week or less (5 treatment days) that can be dosimetrically accounted for in the analysis.
* Negative serum or urine beta-HCG for females of child bearing age.
* Patients will be stratified into 2 groups for evaluation of secondary objective endpoints based on the absence or presence of metastatic disease.
* Patients may enter this study in specific clinical situations often defined by multimodality protocols that include the use of radiation therapy, including irradiation alone or combined with surgery (following surgical resection that may be macroscopically complete or incomplete, with positive or negative histologic margins) and/or chemotherapy (following neoadjuvant chemotherapy or combined with post-irradiation adjuvant chemotherapy).Patients requiring regional nodal irradiation and/or metastatic site irradiation are allowed as long as the primary site requires radiation.Patients with recurrent tumors or second malignant neoplasms are allowed on this study if the current primary tumor site requiring irradiation has not previously been irradiated. The treatment plan detailed in this study will allow most patients to be concurrently enrolled on institutional and COG studies.
* Patients enrolled prior to amendment 4.0, who are still in active participation will be reconsented to the current version of the protocol (5.0).

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 202 (Actual)
Dates: Start 2003-01-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2029-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krasin, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Hua C, Gray JM, Merchant TE, Kun LE, Krasin MJ. Treatment planning and delivery of external beam radiotherapy for pediatric sarcoma: the St. Jude Children's Research Hospital experience. Int J Radiat Oncol Biol Phys. 2008 Apr 1;70(5):1598-606. doi: 10.1016/j.ijrobp.2007.12.013. Epub 2008 Jan 30. PMID 18234441
- [Background] Krasin MJ, Davidoff AM, Xiong X, Wu S, Hua CH, Navid F, Rodriguez-Galindo C, Rao BN, Hoth KA, Neel MD, Merchant TE, Kun LE, Spunt SL. Preliminary results from a prospective study using limited margin radiotherapy in pediatric and young adult patients with high-grade nonrhabdomyosarcoma soft-tissue sarcoma. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):874-8. doi: 10.1016/j.ijrobp.2009.02.074. Epub 2009 Jul 20. PMID 19625137
- [Background] Krasin MJ, Xiong X, Reddick WE, Ogg RJ, Hoffer FA, McCarville B, Kaste SC, Spunt SL, Navid F, Davidoff AM, Zhang L, Kun LE, Merchant TE. A model for quantitative changes in the magnetic resonance parameters of muscle in children after therapeutic irradiation. Magn Reson Imaging. 2006 Dec;24(10):1319-24. doi: 10.1016/j.mri.2006.08.004. Epub 2006 Oct 25. PMID 17145403
- [Background] Hua C, Shukla HI, Merchant TE, Krasin MJ. Estimating differences in volumetric flat bone growth in pediatric patients by radiation treatment method. Int J Radiat Oncol Biol Phys. 2007 Feb 1;67(2):552-8. doi: 10.1016/j.ijrobp.2006.08.069. Epub 2006 Nov 9. PMID 17097831
- [Background] M.J. Krasin; X. Xiong; L. Zhang; W.E. Reddick; T.E. Merchant. A Prospective Study of Quantitative Changes in the Musculature of Children Treated with Radiation Therapy for Sarcomas International journal of radiation oncology, biology, physics(volume 63 issue Pages S443-S444), 2005
- [Background] Krasin, M J; T.E. Merchant; S.L. Spunt; A.M. Davidoff; F. Navid; S. Wu; X. Xiong; C. Hua; L.E. Kun Early Results of a Prospective Study Delivering Limited Margin Radiotherapy for Pediatric Non-Rhabdo-Soft Tissue Sarcomas (NRSTS) and Aggressive Fibromatoses (AF) International journal of radiation oncology, biology, physics(volume 66 issue 3 Page S112), 2006
- [Background] Krasin MJ, MD; Xiong X, PhD; Hua C, PhD; Marchese VG, PT, PhD; Cremer L, PT; Zhang L; Spunt SL, MD; Navid F, MD; Merchant TE, DO,PhD. A Model for Changes in Jaw Function in Children Following Therapeutic Irradiation of the Head and Neck presented at The 9th International Conference on Long-term Complications of Treatment of Children and Adolescents for Cancer, 2006
- [Derived] Tinkle CL, Pappo A, Wu J, Mao S, Hua CH, Shulkin BL, McCarville MB, Kaste SC, Davidoff AM, Bahrami A, Green DM, Ness KK, Merchant TE, Spunt SL, Krasin MJ. Efficacy and Safety of Limited-Margin Conformal Radiation Therapy for Pediatric Rhabdomyosarcoma: Long-Term Results of a Phase 2 Study. Int J Radiat Oncol Biol Phys. 2020 May 1;107(1):172-180. doi: 10.1016/j.ijrobp.2020.01.011. Epub 2020 Jan 25. PMID 31987969
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 202 participants were enrolled between January 10, 2003 and July, 9, 2014.
Pre-assignment Details: A total of 202 patients were enrolled in the study. Of 202 patients, 167 patients completed the study requirements, progression, death, and secondary malignancy, 9 patients still are in follow-up, and 26 patients were off study early due to parent or patient request, PI discretion, physician's discretion, Ineligible, and not returning to St. Jude. Completed ACT trial.
Groups:
- Treatment: Eligible patients will be accessioned at the time of irradiation and undergo a pre-radiotherapy evaluation, treatment planning, image-guided radiotherapy delivery and intra-and post-irradiation evaluations.
  image-guided radiotherapy: Conformal limited image radiotherapy is radiation therapy that targets tumors with a prescribed dose of radiation which allows the surrounding normal tissues to remain basically untreated.
  A total of 202 patients were enrolled in the study. Of 202 patients, 167 patients completed the study requirements, progression, death, and secondary malignancy, 9 patients still are in follow-up, and 26 patients were off study early due to parent or patient request, PI discretion, physician's discretion, Ineligible, and not returning to St. Jude. Completed ACT trial.
Period: Overall Study
Arm/Group | Treatment
Started | 202
Completed | 167
Not Completed | 35
Not completed — Withdrawal by Subject | 5
Not completed — Physician's discretion | 13
Not completed — PI Discretion | 4
Not completed — Ineligible | 2
Not completed — Lost to Follow-up | 2
Not completed — Still on Study | 9

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.84 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 190
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 45
  Black and White | 2
  Other | 3
  Unknown | 1
  White | 151

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Local Failures at 5 Years in Patients With Image Guided Radiation Therapy
Description: The cumulative incidence of local failures is used to report the control of local failures in patients with image guided radiation therapy as defined in this study for patients with primary musculoskeletal tumors (MST).
Time Frame: 5-years follow-up after completion of therapy.
Population: Of 202 patients enrolled in the study, 199 patients were treated with radiation therapy. Three patients were off study before radiation therapy. Cumulative incidence of local failure is calculated from completion of RT to dates of local failure, distant failure (metastatic), the secondary malignancy, death, or off study (last contact) while distant failure (metastatic), the secondary malignancy, and death are considered as competing risks.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Treatment: Eligible patients will be accessioned at the time of irradiation and undergo a pre-radiotherapy evaluation, treatment planning, image-guided radiotherapy delivery and intra- and post-irradiation evaluations. Conformal limited image radiotherapy is radiation therapy that targets tumors with a prescribed dose of radiation which allows the surrounding normal tissues to remain basically untreated.
Arm/Group | Treatment
Number analyzed (Participants) | 199
percentage of patients | 13.37 [9.02 to 18.57]

2. Primary Outcome: Cumulative Incidence of Local Failures at 10 Years in Patients With Image Guided Radiation Therapy
Description: as for outcome 1
Time Frame: 10- years follow-up after completion of therapy
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 199
percentage of patients | 14.31 [9.68 to 19.81]

3. Secondary Outcome: Changes in Growth Rate and Length of Bone, Bone Density, Development of Muscle (Muscle Function, e.g. Range of Motion), Occurrence of Organ Specific (e.g. Lung, Skin) CTC Measured Toxicities.
Description: Investigate the dose and volume relationship for the developing physis and cortical bone using physical measures and imaging evaluations.
Time Frame: Time to local failure (local control) over 5 years follow-up after completion of therapy
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Growth Rate and Length of Bone, Bone Density, Development of Muscle (Muscle Function, e.g. Range of Motion), Occurrence of Organ Specific (e.g. Lung, Skin) CTC Measured Toxicities.
Description: as for outcome 3
Time Frame: Time to local failure (local control) over 10 years follow-up after completion of therapy
Reporting Status: Not Posted

5. Secondary Outcome: Muscle Function Over Time, PET, DCE-MR, T2* MR Quantitative Parameters.
Description: Describe the severity and time course of radiation-induced changes in the soft tissues and adjacent organs, including muscle and subcutaneous tissues.
Time Frame: Change from baseline as well as comparison to non-treated side (when available) during the first 5 years after completion of therapy.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events collected from the time of enrollment out to 10 years or 18 years of age post treatment.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 2/199
Serious Adverse Events (participants affected / at risk) | 9/199
Other Adverse Events (participants affected / at risk) | 50/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=199)
Middle ear/hearing (Ear and labyrinth disorders) | 1 (1)
Wound-infectious (Skin and subcutaneous tissue disorders) | 2 (2)
Hepatic-Other (Hepatobiliary disorders) | 1 (1)
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 1 (1)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=199)
Weight loss (General disorders) | 1 (1)
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 2 (2)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 14 (15)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Gastrointestinal-Other (Gastrointestinal disorders) | 1 (1)
Mucositis due to radiation (Gastrointestinal disorders) | 4 (4)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 2 (2)
Melena/GI bleeding (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin (Infections and infestations) | 1 (1)
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 4 (4)
Syncope (Nervous system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Keratitis (corneal inflammation/corneal ulceration (Eye disorders) | 1 (1)
Ocular-Other (Eye disorders) | 1 (2)
Headache (General disorders) | 1 (1)
Pain due to radiation (General disorders) | 2 (2)
Pain due to radiation, 900180 (General disorders) | 5 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/Genitourinary-Other (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Sexual/Reproductive Function-Other (Reproductive system and breast disorders) | 1 (1)
Syndromes-Other (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT00186992/Prot_SAP_000.pdf